CLINICAL TRIAL: NCT07399509
Title: Prospective Observational Study Evaluating the Sexual Function After Insertion of an Artificial Urinary Sphincter in Women
Brief Title: Evaluation of Sexual Function After Artificial Urinary Sphincter Implantation
Acronym: SPHINCTER
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251272; 2025-A01903-46 (Other: IDRCB)
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Female Artificial Urinary Sphincter Implantation
Keywords: Artificial urinary sphincter; Urinary Incontinence; Sexual function; Sexual quality of life
MeSH Terms: conditions — Urinary Incontinence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — The PISQ-12 questionnaire, which explores female sexual function; the ICIQ-FLUTSsex questionnaire, which focuses on the impact of urinary leakage on sexuality; the USP questionnaire, which assesses the frequency and characteristics of urinary incontinence; and the Qualiveen-SF questionnaire, which measures the impact of these urinary disorders on daily life. A bladder diary was completed preoperatively as well as during follow-up visits at 6 and 12 months.

SUMMARY:
Urinary incontinence (UI) is a common and disabling condition that affects millions of people worldwide and significantly impacts the quality of life of those affected. It is well established that urinary incontinence negatively affects sexual life. Although there is no definitive consensus yet, many authors report that sexual function, after surgical intervention to restore continence, is likely to improve or, at the very least, remain unchanged.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate sexual function in women 6 months after implantation of an artificial urinary sphincter.

Patients will be informed during the preoperative consultation, with an information sheet provided. Consent to non-opposition will be collected either during the preoperative consultation or on the day of the procedure, if additional time for reflection is needed. Questionnaires will be completed during follow-up visits at 6 and 12 months postoperatively.

The patients concerned are women who have undergone implantation of an artificial urinary sphincter.

Patients will be informed during the preoperative consultation, with an information sheet provided. Consent to non-opposition will be collected either during the preoperative consultation or on the day of the procedure, if additional time for reflection is needed. Questionnaires will be completed during follow-up visits at 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 80 years
* Patients with from urinary incontinence with an appropriate surgical indication for artificial urinary sphincter implantation
* Patients who accept the surgical indication and have signed the informed consent for the procedure
* No objection from the patients to participate in the study after reading the information sheet

Exclusion Criteria:

* - Pregnant or breastfeeding patients
* Life expectancy of less than 2 years
* Patients who have undergone colpocleisis surgery
* Patients with neurological conditions causing loss of sensation
* Patients reporting no interest in sexual activity
* Patients suffering from chronic pelvic pain

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients who have benefited from the surgical implantation of an artificial urinary sphincter
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Assess sexual function | 6 months
  sexual quality of life assessed at 6 months post operatively by the PISQ-12 questionnaire (scale from 0 to 48).

SECONDARY OUTCOMES:
Assess sexual function | 12 months
  sexual quality of life assessed at 12 months post operatively by the PISQ-12 questionnaire.
Assess sexual quality of life | 6 and 12 months
  sexual quality of life assessed at 6 and 12 months post operatively by the ICIQ-FLUTSsex questionnaire.
Assess urinary incontinence (clinical efficacy) | 6 and 12 months
  sexual quality of life assessed at 6 and 12 months post operatively by the USP questionnaire.
Assess urinary incontinence (clinical efficacy) | 6 and 12 months
  A voiding diary at 6 and 12 months (reporting the number of leaks per day),with a comparison to the preoperative value. Where applicable, the number of pads used per day.
Assess quality of life | 6 and 12 months
  Quality of life assessed at 6 and 12 months post operatively by the Qualiveen SF questionnaire.
Assess complications | 6 and 12 months
  Surgical complications assessed at 6 and 12 months post according to the Calvien Dindo.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique PHE, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, service d'urologie, Paris, France

IPD SHARING:
Plan to Share IPD: No